CLINICAL TRIAL: NCT04065802
Title: Stereotactic Arrhythmia Radioablation for Ventricular Tachycardia Management
Acronym: STAR VTM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Calgary (Other)
Collaborators: Libin Cardiovascular Institute of Alberta (Other)
Responsible Party: Principal Investigator, Vikas Kuriachan, Clinical Associate Professor (Cardiology/EP), University of Calgary
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REB19-1281
Record Dates: First submitted 2019-08-20; First posted 2019-08-22 (Actual); Last update posted 2022-11-15 (Actual); Status verified 2022-11

CONDITIONS: Stereotactic Radioablation for Ventricular Tachycardia

STUDY DESIGN:
Intervention Model Description: Adult patients with a cardiomyopathy and ventricular tachycardia who have failed conventional anti-arrhythmic management.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Radioablation Treatment (Experimental): Patients will receive radioablation to scar regions of the heart responsible for ventricular tachycardia
  Interventions: Radiation: Stereotactic Radioablation

INTERVENTIONS:
Radiation: Stereotactic Radioablation — External, non-invasive radiation delivery to scar regions of heart to treat ventricular arrhythmias

SUMMARY:
Stereotactic Arrhythmia Radioablation (STAR) ablation is a safe and feasible option for cardiomyopathy patients for management of refractory ventricular tachycardia.

STAR can be performed with available cardiac imaging, prior mapping/electrogram information, and standard ECGs without a multi-electrode ECG vest.

DETAILED DESCRIPTION:
Study Hypotheses:

1. Stereotactic Arrhythmia Radioablation (STAR) ablation is a safe and feasible option for cardiomyopathy patients for management of refractory ventricular tachycardia.
2. STAR can be performed with available cardiac imaging, prior mapping/electrogram information, and standard ECGs without a multi-electrode ECG vest.

Study Objectives:

1. Evaluate the safety of STAR in a local cohort
2. Estimate effectiveness of STAR in reducing VT burden

Study Design: Prospective single center, single arm, non-randomized trial.

Number of patients: 20 patients

Study Duration: Enrollment will occur over three years and at least minimum follow up of six months

Study Population: Adult patients with a cardiomyopathy and ventricular tachycardia who have failed conventional anti-arrhythmic management.

Primary safety endpoint: Any treatment-related serious adverse events in the first 90 days.

Primary efficacy endpoint: Reduction in VT episodes tracked by ICD with a six week blanking period.

Statistical methodology: Wilcoxon matched-pairs signed-ranks test to compare the number of treated episodes before and after.

Assessment of events: Adjudicated by study investigators

Economic Analysis: Costs and resources required for STAR .Compare costs between the patients undergoing STAR with conventional catheter-based VT ablation.

ELIGIBILITY:
Inclusion Criteria:

18 years of age and have an implanted cardioverter defibrillator (ICD) with:

1. Structural heart disease: ischemic or non-ischemic cardiomyopathy diagnosed with cardiac imaging demonstrating either segmental myocardial dysfunction, or presence of scar.
2. At least one of the following monomorphic VT events despite prior attempted catheter ablation (or contraindication for ablation), and despite treatment with a class III antiarrhythmic drug (contraindicated, ineffective or not tolerated):

A: Sustained monomorphic VT documented on 12-lead ECG or rhythm strip terminated by pharmacologic means, DC cardioversion or manual ICD Therapy.

B: ≥3 episodes of monomorphic VT treated with antitachycardia pacing (ATP), at least one of which was symptomatic C: ≥ 5 episodes of monomorphic VT treated with antitachycardia pacing (ATP) regardless of symptoms D: ≥1 appropriate ICD shocks, E: ≥3 monomorphic VT episodes within 24 hours VT events must be confirmed by ECG/monitor or ICD download.

Exclusion Criteria:

* Has received prior radiotherapy to the anticipated treatment field
* Pregnancy
* Unable to unwilling to provide informed consent
* New York Heart Association class IV heart failure or inotrope use limiting the safe transport to the radiotherapy suite
* Patients in whom the only ventricular arrhythmias are ventricular fibrillation, torsade de pointes, or polymorphic ventricular tachycardia.
* Active coronary ischemia in the last 30 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-04-14 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Efficacy of radiation treatment for VT reduction | 6 month period before treatment to the 6 month period after ablation with a 6 week blanking period post-treatment.
  Reduction in VT burden tracked by ICD and defined as the difference between the number of ICD-treated VT/VF episodes comparing the 6 months prior to treatment to the 6 months after treatment.
Safety composite endpoint of radiation treatment-related pericarditis, pneumonitis, changes in cardiac structures, function, and/or ICD function. | 90 days after treatment
  Any treatment-related serious adverse events including pericarditis, radiation pneumonitis, deterioration in cardiac function, new or worsening cardiac valve dysfunction, and implantable cardioverter defibrillator malfunction.

SECONDARY OUTCOMES:
Overall mortality | Six months
  Six month survival after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Vikas Kuriachan, MD, Principal Investigator — University of Calgary
Locations (1):
- University of Calgary, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No
The data will be anonymous. Given the small number of patients in the study individual treatments and outcomes maybe looked at.

REFERENCES:
- [Result] Cuculich PS, Schill MR, Kashani R, Mutic S, Lang A, Cooper D, Faddis M, Gleva M, Noheria A, Smith TW, Hallahan D, Rudy Y, Robinson CG. Noninvasive Cardiac Radiation for Ablation of Ventricular Tachycardia. N Engl J Med. 2017 Dec 14;377(24):2325-2336. doi: 10.1056/NEJMoa1613773. PMID 29236642
- [Result] Cuculich PS, Robinson CG. Noninvasive Ablation of Ventricular Tachycardia. N Engl J Med. 2018 Apr 26;378(17):1651-1652. doi: 10.1056/NEJMc1802625. No abstract available. PMID 29694814